CLINICAL TRIAL: NCT00253266
Title: Comparison of Venlafaxine Augmentation With Quetiapine v.s. Placebo in Treatment Resistant Depression
Brief Title: Venlafaxine Augmentation in Treatment Resistant Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01/2005; 2005-001217-17 (EudraCT Number)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Depression
Keywords: Treatment resistant depression; Augmentation; Pharmacogenetics
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant | interventions — Venlafaxine Hydrochloride; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verum (Experimental): Quetiapine augmentation
  Interventions: Drug: Venlafaxine; Drug: Quetiapine
- Placebo (Placebo Comparator): "Placebo" augmentation
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Venlafaxine — Venlafaxine XR up to 450 mg/d during the complete trial (8 weeks)
  Other Names: Trevilor retard
Drug: Quetiapine — Quetiapine up to 200 mg/d for four weeks
  Other Names: Seroquel
  Arms: Verum

SUMMARY:
This is an assessment of the efficacy of venlafaxine-HCL augmentation with the neuroleptic quetiapine in treatment resistant depression.

DETAILED DESCRIPTION:
We examine the efficacy of Venlafaxine-HCL augmentation with the neuroleptic Quetiapine in treatment resistant depression in a double-blind randomized clinical trial. Secondary objective is the evaluation of pharmacogenetic factors contributing to drug efficacy in treatment resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* Female and male inpatients with a major depressive disorder without psychotic features or with a depressive episode within a bipolar I or II disorder without psychotic features
* Ages between 20 and 70 years
* Total score greater than 18 on the Hamilton Depression Rating Scale
* Documentation of at least one ineffective antidepressant drug trial under adequate dosage for at least 6 weeks in the current episode

Exclusion Criteria:

* Other psychiatric axis I disorders than those mentioned as Inclusion criteria
* Acute suicidality (Item 3 of the Hamilton Depression Rating Scale greater than 2)
* Drug or alcohol addiction
* Patients with severe hepatic, cardiovascular, neurologic, metabolic or malignant disorders
* Documentation or report of a previous ineffective treatment trial with venlafaxine, lamotrigine or quetiapine
* Functional kidney disorders
* Untreated hypertension
* Acute treatment with thyroid hormone (less than 3 months)
* Pregnant or nursing patients
* Women of childbearing age without effective contraception

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-04; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | after monotherapy and after augmentation

SECONDARY OUTCOMES:
Self reported psychopathology (Beck Depression Inventory [BDI], State-Trait Anxiety Inventory [STAI]) | after monotherapy and after augmentation
Cognitive function | after monotherapy and after augmentation

CONTACTS AND LOCATIONS:
Overall Officials: Florian Holsboer, MD, PhD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Bavaria, Germany